CLINICAL TRIAL: NCT05145478
Title: CTA_IIT_CRUSH PAD: Real-world Outcomes Following Use of the Shockwave Intravascular Lithotripsy (IVL) Technology in Calcified Common Femoral Lesions
Brief Title: CRUSH PAD: Real-world Outcomes Following Use of Shockwave Intravascular Lithotripsy (IVL) Technology in Calcified Common Femoral Lesions
Status: Recruiting | Type: Observational
Sponsor: Yale University (Other)
Collaborators: Shockwave Medical, Inc. (Industry); Brown University (Other)
Responsible Party: Sponsor
Other Study IDs: 2000031113
Record Dates: First submitted 2021-11-15; First posted 2021-12-06 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Femoral Arterial Calcification; Peripheral Arterial Disease; Claudication; Critical Limb Ischemia
Keywords: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Shockwave Intravascular Lithotripsy (IVL): Patients with calcified common-femoral artery disease, who are eligible to receive IVL per the FDA indications.
  Interventions: Device: Shockwave Intravascular Lithotripsy (IVL)

INTERVENTIONS:
Device: Shockwave Intravascular Lithotripsy (IVL) — Eligible patients with atherosclerotic lesions in the femoral artery who either have claudication or critical limb ischemia will receive endovascular treatment in addition to be treated with Shockwave Intravascular Lithotripsy (IVL) technology.

SUMMARY:
The primary goal of the study is to obtain effect size data on the use of Shockwave Intravascular Lithotripsy (IVL) technology in calcified common femoral lesions in patients with peripheral artery disease for a series of endpoints, including target lesion revascularization and health status, to enable future planning of comparative effectiveness research.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the generic health status outcomes and efficacy and safety outcomes following use of the Shockwave Intravascular Lithotripsy (IVL) technology in calcified common femoral lesions in patients with PAD seen in routine clinical practice.

The main testable hypothesis is that the use of IVL is associated with a health status improvement that is equal or higher than the threshold of a minimally clinically important difference on the EQ5D. Preliminarily data will be derived for the primary endpoint target lesion revascularization to enable future planning of larger comparative effectiveness research.

Secondary objectives of the study are to document procedural success following the use of IVL in common femoral lesions, disease stage change, as well as disease-specific health status in the real-world.

ELIGIBILITY:
Inclusion Criteria:

* Subjects presenting with claudication or CLI by Rutherford Clinical Category 2, 3, 4, 5, or 6 of the target limbs
* Subject is a suitable candidate for angiography and endovascular intervention per the latest clinical guidelines
* Patient is scheduled to undergo treatment with Shockwave Intravascular Lithotripsy (IVL) technology followed by standard of care treatment with DCB, BMS, DES at the physician's discretion.

Angiographic Inclusion Criteria

* Target lesion that is located in a native, de novo common femoral artery
* Target lesion reference vessel diameter is between 4.0mm and 7.0mm by visual estimate.
* Target lesion is ≥70% stenosis by investigator via visual estimate.
* Target lesion length is ≤50mm for lesions 70-99% stenosed. Target lesion can be all or part of the 50mm treated zone.
* Chronic total occlusion, lesion length is ≤50mm of the total ≤50 mm target lesion.
* Calcification is at least moderate defined as presence of fluoroscopic evidence of calcification: 1) on parallel sides of the vessel and 2) extending > 50% the length of the lesion if lesion is ≥50mm in length; or extending for minimum of 20mm if lesion is <50mm in length.

Exclusion Criteria:

* Subjects with any medical condition that would make him/her an inappropriate candidate for treatment with Shockwave Medical Peripheral Lithoplasty® System as per Instructions for Use (IFU) or investigator's opinion.
* Subject is already enrolled in other investigational (interventional) studies that would interfere with study endpoints.
* Cognitive impairment as documented in medical records
* Not speaking English or Spanish
* Currently a prisoner
* Pregnancy or nursing
* Estimated survival less than 12 months at the time of screening
* Prior history of CFA endarterectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population include patients with atherosclerotic lesions in the femoral artery who either have claudication or critical limb ischemia who are eligible to receive endovascular treatment in addition to be treated with Shockwave Intravascular Lithotripsy (IVL) technology.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in Generic Health Status | Baseline and 30 days
  Generic Health Status will be measured using the EQ5D health status assessment. Descriptive system for health-related quality of life states in adults, consisting of five dimensions (Mobility, Self-care, Usual activities, Pain & discomfort, Anxiety & depression), each of which has five severity levels that are described by statements appropriate to that dimension. Higher scores indicate more severe or frequent problems.
Change in Generic Health Status | Baseline and 6 months
  Generic Health Status will be measured using the EQ5D health status assessment. Descriptive system for health-related quality of life states in adults, consisting of five dimensions (Mobility, Self-care, Usual activities, Pain & discomfort, Anxiety & depression), each of which has five severity levels that are described by statements appropriate to that dimension. Higher scores indicate more severe or frequent problems.
Rate of Procedural Success | Immediately post procedure
  Procedural success defined as residual stenosis ≤30% without flow-limiting dissection (≥ grade D) prior to DCB

SECONDARY OUTCOMES:
Number of Patients Free from TLR | Up to 12 months
  Freedom from clinically driven target lesion revascularization (TLR). Assessed at 30 days, 6 months and 12 months.
Number of patients with new-onset MAEs | Up to 12 months
  The composite of new-onset Major Adverse Events (MAEs) is comprised of:
  * Need for emergency surgical revascularization of target limb, including CFA endarterectomy
  * Unplanned target limb major amputation (above the ankle)
  * Symptomatic thrombus or distal emboli that require surgical, mechanical, or pharmacologic means to improve flow and extend hospitalization
  * Perforations that require an intervention, including bail-out stenting
Rate of Periprocedural clinical success | During admission, before discharge up to 48 hours
  Periprocedural clinical success as defined by residual stenosis ≤30% without flow-limiting dissection (≥ grade D) prior to DCB or stenting.
Change in Clinical Success | Baseline and 30 days
  Rutherford Category. Classification of PAD into acute and chronic limb ischemia associated by clinical symptoms. Evaluates patient's chronic limb pain and claudication by ABI/TBI. The category scale is from 0-6. The clinical interpretation of the scale is that a higher category indicates a worse condition.
Change in Clinical Success | Baseline, 6 months and 12 months
  Rutherford Category. Classification of PAD into acute and chronic limb ischemia associated by clinical symptoms. Evaluates patient's chronic limb pain and claudication by ABI/TBI. The category scale is from 0-6. The clinical interpretation of the scale is that a higher category indicates a worse condition.

OTHER OUTCOMES:
Change in Health Status | Baseline, 30 days and 6 months
  Health status will be measured using the disease-specific Peripheral Artery Questionnaire (PAQ). PAD-specific, multi-dimensional health status instrument with a CLI specific module. Higher scores indicate better functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Mena-Hurtado, MD, Principal Investigator — Yale University; Kim Smolderen, PhD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale New Haven Health, New Haven, Connecticut
  - The Miriam Hospital, Providence, Rhode Island